CLINICAL TRIAL: NCT00980616
Title: Effect of the Injection of Local Analgesia With Epinephrine During Total Hip Arthroplasty on the Blood Losses Per and Operatively.
Brief Title: Use of Local Analgesia With Epinephrine During Total Hip Arthroplasty (THA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0056
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Arthroplasty, hip; blood losses; pain; local analgesia; epinephrine; Primary total hip arthroplasty
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ropivacaine, serum, adrenalin (Experimental): 235 mg of ropivacaine, 5 ml physical serum and 0.5 mg of adrenalin.
  Interventions: Drug: ropivacaine, physical serum and adrenalin
- No infiltration (No Intervention): B: no infiltration

INTERVENTIONS:
Drug: ropivacaine, physical serum and adrenalin — A: experimental group: 235 mg of ropivacaine, 5 ml physical serum and 0.5 mg of adrenalin
  Arms: Ropivacaine, serum, adrenalin

SUMMARY:
The aim is to determine if the use of infiltration with an adrenalin solution in the operative field of Total Hip Arthroplasty (THA), allays a significant reduction of the cumulated volume of bleeding (pre and post operative) without increasing the per and post operative risks. At the same time, the effect on the post operational pains is evaluated.

DETAILED DESCRIPTION:
This prospective randomized study compares a population receiving a local anaesthetic (ropivacaine, adrenalin and physiological serum) in the operative field to a population undergoing a standard protocol.

The cumulated volume of bleeding per and post operative are recorded and complete blood count (CBC).

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty
* Age between 50 and 85

Exclusion Criteria:

* fracture of the femoral neck
* patients with contraindications for local anaesthesia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
measuring volume of cumulated bleeding per and post operative and analyse of complete blood count (CBC) | pre and post operative

SECONDARY OUTCOMES:
Womac score pre operative, at 3 months and at 12 months | at 3 months and 12 months
Visual analogue pain score (VAS) during hospitalisation | at 3 months and 12 months
Consumption of analgesics | at 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Descamps, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand (orthopaedic surgery), Clermont-Ferrand, France